## THE EFFECT OF HEALTH PROMOTION PROGRAM APPLIED TO UNIVERSITY STUDENTS ON IMPROVING HEALTHY NUTRITION AND PHYSICAL ACTIVITY BEHAVIORS

### INFORMED CONSENT FORM

Date of the Document: January 1, 2019

Primary Investigator: Ayse Dost, Lecturer Istanbul Medipol University Faculy of Health Sciencies Nursing Department Adress: Unkapanı Mah. Atatürk Bulvarı No: 27, 34083 Fatih, İstanbul Phone: 4448544

Sponsor: İstanbul Medipol Üniversitesi Hastanesi Phone: 444 85 44 Fax :0212 521 23 77 Adress: Unkapanı Mah. Atatürk Bulvarı No: 27, 34083 Fatih, İstanbul

We are conducting a research to identify people who will participate in the Health Promotion Program for University Students. We recommend that you participate in this research. Participation in the study is voluntary. If you want to participate after reading the information below, sign the form.

Some measurements will be made to determine your healthy eating and physical activity behaviors and to determine your obesity and cardiovascular risk status. After these measurements, you will be included in the behavior change program, which will last for six months. The same measurements will be made again to reveal the changes that occur at the end of the program.

You will not be charged for participating in this study. You will not be paid for participating in the study.

#### Possible benefits of the research:

This study aims to develop healthy eating and physical activity behaviors.

You may refuse to participate in this study. Participation in this research is entirely voluntary and you have the right to withdraw your consent at any stage of the study.

#### **Student's Declaration**

Mrs. Ayşe Dost stated that a study titled is The Effect of Health Promotion Program Applied to University Students on Improving Healthy Nutrition and Physical Activity Behaviors will be conducted in my university. After this information, I was invited as a participant to such a research.

If I participate in this research, I believe that the confidentiality of the information that I should keep between me and the researcher will be treated with great care and respect during this research. I have been given sufficient confidence that my personal information will be carefully protected during the use of the research results for educational and scientific purposes.

I can withdraw from the research without giving any reason during the execution of the project. (However, I am aware that it would be appropriate to let me know in advance that I will withdraw from the research in order not to leave the researchers in a difficult position). I may also be excluded from the research by the researcher, provided that no harm to my health condition is provided.

I do not assume any monetary responsibility for the expenditures to be made for the research. I will not be paid. I don't have to participate in this research and I may not. I haven't been compelled to participate in the investigation. I also know that if I refuse to participate, it will not cause any harm.

I have understood all the explanations made to me in detail. I decided to take part in this research project as a "participant I am after a certain period of thinking on my own. I accept this invitation with great pleasure and volunteering.

I will receive a copy of this signed form.

# Participant Name and surname:

Address: Wire. Signature

## **Interview witness Name and surname:**

Address: Wire. Signature:

Researcher interviewing the participant: Ayse Dost, Lecturer

Address: Istanbul Medipol University Faculy of Health Sciencies Nursing Department

Unkapanı Mah. Atatürk Bulvarı No: 27, 34083 Fatih, İstanbul

Phone: 4448544

Signature: